CLINICAL TRIAL: NCT05963230
Title: ScanNav Anatomy PNB FDA Data Collection Plan
Status: Completed | Type: Observational
Sponsor: IntelligentUltrasound Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: IU2023_AG_12
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Ultrasound Recordings

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Volunteer Participants: Healthy adult (18+ years old) volunteers
  Interventions: Other: Ultrasound scans

INTERVENTIONS:
Other: Ultrasound scans — Ultrasound scans collected by experts in ultrasound-guided regional anaesthesia.

SUMMARY:
To gather additional training and/or validation data (recorded ultrasound scans) for ScanNav Anatomy PNB in the following categories:

* Femoral Nerve (Femoral)
* Interpectoral (PECS I) and pectoserratus (PECS II)
* Transversus abdominis plane (TAP)
* Serratus Plane (SP)
* Infra-inguinal Facia Iliaca (Infra-inguinal FI) Data will be collected in the form of "scenes" (target block view) and "non-scenes" (areas adjacent to the target block view).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age;
* Able to comprehend and sign the Informed Consent prior to enrolment in the study.

Exclusion Criteria:

* Aged <18 years of age;
* Unwilling or unable to provide informed consent.
* Previous history of medical interventions that may affect the anatomy of the chosen scan areas, e.g. hip replacements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers from the San Diego, California, USA region.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Ultrasound scan recordings | 6 months
  Ultrasound scan recordings collected by experts in ultrasound-guided regional anaesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: James Bowness, Dr, Principal Investigator — Intelligent Ultrasound
Locations (1):
- Taylor Research, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No